CLINICAL TRIAL: NCT05959421
Title: Durability of Immunity Induced by the Ebolavirus Vaccine VSV-EBOV and As-sessment of a Booster Dose for Pre-Exposure Prophylaxis in Individuals at Potential Occupational Risk for Ebolavirus Exposure
Brief Title: Immunity Induced by VSV-EBOV and Assessment of a Booster Dose in Individuals at Potential Occupational Risk for Exposure
Acronym: PREPARE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Bernhard Nocht Institute for Tropical Medicine (Other Government); Goethe University (Other); German Federal Ministry of Education and Research (Other Government); Monipol Deutschland GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PREPARE-GERMANY
Record Dates: First submitted 2023-05-21; First posted 2023-07-25 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Ebola Vaccine
Keywords: Ebola, VSV-EBOV, vaccine, immunity
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Intervention Model Description: Randomized non-blinded interventional trial Type of control: Randomized - Booster or no booster at 6 months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Booster (Experimental): Participants will receive ERVEBO® (rVSV∆G-ZEBOV-GP) ≥72 million pfu/mL primary immunization And a single booster immunization with the same dose of study vaccine as the primary dose (≥72 million pfu/mL) at month 6 following primary vaccination
  Interventions: Biological: ERVEBO® (rVSV∆G-ZEBOV-GP)
- no Booster (Experimental): Participants will receive ERVEBO® (rVSV∆G-ZEBOV-GP) ≥72 million pfu/mL primary immunization only
  Interventions: Biological: ERVEBO® (rVSV∆G-ZEBOV-GP)

INTERVENTIONS:
Biological: ERVEBO® (rVSV∆G-ZEBOV-GP) — intramuscular vaccination
Biological: ERVEBO® (rVSV∆G-ZEBOV-GP) — intramuscular vaccination
  Arms: Booster

SUMMARY:
This study is a multi-center, open label, randomized phase 3b trial to assess the durability of Immunity induced by the Ebolavirus Vaccine VSV-EBOV ( with or without booster vaccination) in individuals at potential occupational risk for ebolavirus exposure

DETAILED DESCRIPTION:
All participants will receive a single dose of ERVEBO® (≥72 million pfu) on Day 0. The participants will receive a diary to document local and defined systemic adverse events for 14 days after vaccination. We will collect grade 3 and 4 adverse events after vaccination and at Month 1 and Month 7, and seri-ous adverse events (SAE) for the duration of the study, and assess the immune response at Months 1, 3, 6, 7, 12, 18, 24. In a subgroup (Innate Subgroup) we are also going to assess innate immune response at Day 1 and 3 and Month 6 + Day 1 and Month 6 + Day 3.

A single booster immunization with the same dose as the primary dose (≥72 million pfu/mL) will be given to those randomized to the booster arm of the trial six months after primary vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age ≥18 years.
2. Signed informed consent for the trial.
3. At risk of occupational exposure to Ebola virus through laboratory, clinical contact, or field work, in the judgment of the investigator.
4. Females of child-bearing potential (FOCP) must be willing to use effective methods of con-traception as per the requirements of the protocol (9.3.7) from at least 30 days prior to vac-cination through 2 months following vaccination/booster.
5. Willing to avoid blood and body fluid exposure to high-risk individuals (i.e., immunocompro-mised individuals, individuals receiving immunosuppressive therapy and pregnant or breast-feeding women, children <1 year of age) for at least 6 weeks after vaccination/booster. This includes:

   * Use of effective barrier prophylaxis, such as latex condoms, during any sexual inter-action (regardless of childbearing status or sexual orientation)
   * Avoiding the sharing of needles, razors, eating utensils, drinking from the same cup, or toothbrushes
   * Avoiding open-mouth kissing
   * Use of universal precautions in the health-care setting The investigator can be counseled and may determine when individuals are classified as "immuno-compromised" and what therapy is defined as immunosuppressive therapy in this context.
6. Willing to forgo blood donation 30 days prior to first vaccination until end of study.
7. Willing to accept randomization (boost versus no boost) at month 6 (time window -1 month) visit.

Exclusion Criteria:

1. Any condition that would, in the eyes of the investigator, limit the ability of the participant to meet protocol requirements or would place the participant at unreasonable risk. This includes:

   I) Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health, per the investigator. A clinically significant condition or process includes but is not limited to:
   1. A process that would adversely affect the systemic immune response
   2. A process that would require medication that might adversely affect the systemic immune re-sponse
   3. Any contraindication to repeated injections or blood draws
   4. A condition that requires active medical intervention or monitoring to avert grave danger to the participant's health or well-being during the study period
   5. A condition or process for which signs or symptoms could be confused with reactions to vaccine

   II) Presence of any pre-existing illness or clinical history that, in the opinion of the investigator, would place the participant at an unreasonably increased risk through participation in this study. This in-cludes but is not limited to:
   1. Active malignancy
   2. History of Guillain-Barré Syndrome
   3. History of neurological disorder that may increase risk (history of encephalitis, stroke, or sei-zure)
   4. Active autoimmune disorder requiring systemic immunosuppressive treatment

   III) Any concomitant medication for which reported side effects or adverse events, in the judg-ment of the investigator, may interfere with assessment of safety.

   IV) Participants who, in the judgment of the investigator, will be unlikely or unable to comply with the requirements of this protocol.
2. Pregnant or breast feeding (must have negative pregnancy test on the day of vaccination, prior to vaccination)
3. Known allergy to the components of the rVSV∆G-ZEBOV-GP vaccine (ERVEBO®) vaccine product (VSV, albumin, tris, rice).
4. History of severe local or systemic reactions to any vaccination.
5. Received killed vaccines 14 days before, or intention to receive within 7 days following vac-cination (Day 0)/booster (Month 6).
6. Received live virus vaccines within 30 days before, or intention to receive live virus vaccines within 30 days following, vaccination (Day 0)/booster (Month 6).
7. Received immunoglobulins and/or any blood products within the 120 days preceding vaccina-tion (Day 0)/booster (Month 6).
8. Received allergy treatment with antigen injections within 30 days before vaccination (Day 0)/booster (Month 6).
9. Clinical evidence (e.g. oral temperature >38.0 degrees Celsius, systemic symptoms) of a sys-temic infection or other acute intercurrent illness at the proposed time of vaccination (Day 0)/booster (Month 6).
10. Prior receipt of a vaccine against EVD or prior EVD in medical history.
11. Participation in a clinical trial or use of an investigational product within 30 days or five times the half-life of the investigational product -whichever is longer- prior to receiving the first dose within this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
The course of Anti-EBOV immunoglobulin following primary vaccination | 0-24month
  The course of Anti-EBOV immunoglobulin as measured by EBOV ELISA titers during the 24 months following primary vaccination
Anti-EBOV immunoglobulin at 12 and 24 months follow-up | 12 month follow-up
  Anti-EBOV immunoglobulin as measured by EBOV ELISA titers at 12 and 24 months follow-up
Anti-EBOV immunoglobulin at 12 and 24 months follow-up | 24 month follow-up
  Anti-EBOV immunoglobulin as measured by EBOV ELISA titers at 12 and 24 months follow-up

SECONDARY OUTCOMES:
Occurrence of Grade ≥ 3 AE until one month after primary and booster vaccination | 1 month after primary vaccination
  Number of Grade ≥ 3 AE
Occurrence of Grade ≥ 3 AE until one month after primary and booster vaccination | 1 month after boost vaccination
  Number of Grade ≥ 3 AE
Occurrence of SAE throughout the study | 0-24 month
  Number of serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Marylyn M Addo, Prof, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (2):
- Germany (2):
  - University Hospital Frankfurt (KGU), Frankfurt
  - Bernhard Nocht Centre for Clinical Trials (BNCCT), Hamburg

IPD SHARING:
Plan to Share IPD: No